CLINICAL TRIAL: NCT02027961
Title: A Phase 1 Open-label Study of Safety and Tolerability of MEDI4736 in Subjects With Metastatic or Unresectable Melanoma in Combination With Dabrafenib and Trametinib or With Trametinib Alone
Brief Title: Phase 1 Safety and Tolerability of MEDI4736 in Combination With Dabrafenib and Trametinib or With Trametinib Alone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-ON-MEDI4736-1161
Record Dates: First submitted 2013-11-20; First posted 2014-01-06 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Melanoma
Keywords: Metastatic or Unresectable Melanoma, durvalumab (MEDI4736), dafrafenib, trametinib, BRAF-mutation positive, wild-type BRAF, PD-L1, PD-1
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — durvalumab; dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A1: Durvalumab (3 mg/kg) + Dabrafenib +Trametinib (Experimental): Participants will receive intravenous (IV) dose of 3 milligrams per kilogram (mg/kg) durvalumab every 2 weeks (Q2W) from Day 1 up to 12 months along with oral 150 mg dabrafenib capsule twice daily (BID) and oral 2 mg trametinib tablet once daily (QD) until confirmed disease progression (PD), initiation of alternate cancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue treatment. Post-durvalumab treatment period, participants who developed PD and meet the criteria for re-administration, will receive durvalumab 3 mg/kg up to an additional 12 months and continued the treatment of dabrafenib and trametinib.
  Interventions: Biological: Durvalumab; Drug: Dabrafenib; Drug: Trametinib
- Cohort A2: Durvalumab (10 mg/kg) + Dabrafenib +Trametinib (Experimental): Participants will receive IV dose of 10 mg/kg durvalumab Q2W from Day 1 up to 12 months along with oral doses of dabrafenib 150 mg capsule BID and trametinib 2 mg tablet QD until confirmed PD, initiation of alternate cancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue treatment. Post-durvalumab treatment period, participants who developed PD and meet the criteria for re-administration, will receive durvalumab 10 mg/kg up to an additional 12 months and continued the treatment of dabrafenib and trametinib.
  Interventions: Biological: Durvalumab; Drug: Dabrafenib; Drug: Trametinib
- Cohort B: Durvalumab (10 mg/kg) +Trametinib (Concurrent) (Experimental): Participants will receive concurrent doses of IV 10 mg/kg durvalumab Q2W from Day 1 up to 12 months along with oral dose of trametinib 2 mg tablet QD until confirmed PD, initiation of alternate cancer therapy, unacceptable toxicity, withdrawal of consent, or other reasons to discontinue treatment. Post-durvalumab treatment period, participants who developed PD and meet the criteria for re-administration, will receive durvalumab 10 mg/kg up to an additional 12 months and continued the treatment of trametinib.
  Interventions: Biological: Durvalumab; Drug: Trametinib
- Cohort C: Durvalumab (10 mg/kg) +Trametinib (Sequential) (Experimental): Participants will receive sequential doses of oral trametinib tablet 2 mg QD from Day 1 to Day 42 and IV durvalumab 10 mg/kg Q2W starting from Day 29 (Week 5) up to 12 months. Post-durvalumab treatment period, participants who developed PD and meet the criteria for re-administration, will receive durvalumab 10 mg/kg up to an additional 12 months.
  Interventions: Biological: Durvalumab; Drug: Trametinib

INTERVENTIONS:
Biological: Durvalumab — Intravenous dose of 3 or 10 mg/kg durvalumab.
Drug: Dabrafenib — Oral dose of 150 mg dabrafenib capsule.
  Arms: Cohort A1: Durvalumab (3 mg/kg) + Dabrafenib +Trametinib; Cohort A2: Durvalumab (10 mg/kg) + Dabrafenib +Trametinib
Drug: Trametinib — Oral dose of 2 mg trametinib tablet.

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and characterize the safety profile of durvalumab (MEDI4736) in combination with dabrafenib and trametinib or with trametinib alone in participants with metastatic or unresectable melanoma with BRAF-mutation positive or wild-type (WT) BRAF, respectively.

DETAILED DESCRIPTION:
This is a multicenter, open-label study with a dose escalation phase followed by an expansion phase of durvalumab administered in combination with dabrafenib and trametinib or with trametinib alone in participants with BRAF V600 mutation-positive and WT unresectable or metastatic melanoma, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults >= 18 years old
* Histologically confirmed cutaneous melanoma that is either Stage IIIc (unresectable) or Stage IV (metastatic) and determined to be BRAF V600E or V600K mutation-positive (cohort A) or mutation-negative (cohorts B and C)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease by radiographic or physical examination
* Adequate organ and marrow function
* Willingness to provide consent for biopsies positive or BRAF WT measurable disease and adequate organ and marrow function

Exclusion Criteria:

* Prior treatment with a BRAF inhibitor or MEK inhibitor
* Any prior Grade >= 3 immune-related adverse event while receiving immunotherapy
* Active or prior documented autoimmune disease within the past 2 years
* History of or current risk for retinal vein occlusion (RVO) or central serous retinopathy (CSR)
* History of or current cardiovascular risk including myocardial infarction, >= Class II congestive heart failure, uncontrolled arrhythmias, or refractory hypertension
* Active, untreated central nervous system (CNS) metastases
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2018-04-24 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Dose Limiting Toxicities (DLTs) | From first dose of study drug (Day 1) until the planned 3rd dose of durvalumab (Day 29)
  Dose limiting toxicities are defined as any Grade 3 or higher treatment-related (related to any study drug) toxicity that occurs during the DLT evaluation period. Number of participants with DLTs are reported.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | From first dose of study drug (Day 1) up to 90 days after the last dose (up to 4.5 years)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event is any AE that resulted in death, life threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, is a congenital anomaly/birth defect in offspring of a study participant, is an important medical event that may jeopardize the participant or may require medical intervention. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Abnormal Vital Signs and Physical Examinations Reported as TEAEs | From first dose of study drug (Day 1) up to 90 days after the last dose (up to 4.5 years)
  Number of participants with abnormal vital signs and physical examinations reported as TEAEs are reported.
Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs | From first dose of study drug (Day 1) up to 90 days after the last dose (up to 4.5 years)
  Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported.
Number of Participants With Abnormal Electrocardiograms (ECGs) and Echocardiograms (ECHOs) Reported as TEAEs | From first dose of study drug (Day 1) up to 90 days after the last dose (up to 4.5 years)
  Number of participants with abnormal electrocardiograms (ECGs) and echocardiograms (ECHOs) reported as TEAEs are reported.

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response (OR) | From the first dose of study drug until last participant completes 12 months of treatment (assessed up to 4.5 years)
  Objective Response is defined as confirmed complete response (CR) or confirmed partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1). A confirmed CR is defined as two CRs that were separated by at least 28 days. A confirmed PR is defined as two PRs or an un-confirmed PR and an un-confirmed CR that were separated by at least 28 days. A CR is defined as disappearance of all target and non-target lesions, normalization of tumor marker level and any pathological lymph nodes selected as target lesions must have a reduction in short axis to less than 10 mm. A PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Duration of Response (DOR) | From the first dose of study drug until last participant completes 12 months of treatment (assessed up to 4.5 years)
  Duration of response: Duration from first documentation of OR to first documented PD or death due to any cause, whichever occurs first. CR: disappearance of all target and non-target lesions, normalization of tumor marker level and any pathological lymph nodes selected as target lesions must have a reduction in short axis to less than 10 mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of >= 5 mm, taking as reference smallest sum of diameters since treatment started including baseline sum of diameters.
Progression-free Survival (PFS) | From the first dose of study drug until last participant completes 12 months of treatment (assessed up to 4.5 years)
  Progression-free Survival is defined as duration from the start of treatment with study drug until the first documented PD or death, whichever comes first. PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of >= 5 mm, taking as reference smallest sum of diameters since treatment started including baseline sum of diameters. For participants who are alive and progression-free at the time of data cut-off for analysis, PFS was to be censored at the last tumor assessment date.
Overall Survival | From the first dose of study drug until last participant completes 12 months of treatment (assessed up to 4.5 years)
  Overall survival (OS) is measured from the start of treatment until death. For participants who are alive at the end of study or lost to follow-up, OS was censored on the last date when participants are known to be alive.
Percentage of Participants With Disease Control | From the first dose of study drug until last participant completes 12 months of treatment (assessed up to 4.5 years)
  Disease control is defined as confirmed CR or PR, or stable disease (SD) that was maintained for >= 12 weeks based on RECIST v1.1. A confirmed CR is defined as two CRs that were separated by at least 28 days. A confirmed PR is defined as two PRs or an un-confirmed PR and an un-confirmed CR that were separated by at least 28 days. CR: disappearance of all target and non-target lesions, normalization of tumor marker level and any pathological lymph nodes selected as target lesions must have a reduction in short axis to less than 10 mm. A PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. A SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of diameters while on study.
Maximum Observed Plasma Concentration after First Dose (Cmax, 1st) of Durvalumab | Cohorts A and B: End of infusion on Day 1; Cohort C: End of infusion on Day 29
  Maximum observed plasma concentration of durvalumab after first dose is reported.
Maximum Observed Plasma Concentration at Steady State (Cmax, ss) of Durvalumab | Cohorts A and B: end of infusion on Day 141; Cohort C: end of infusion on Day 169
  Maximum observed plasma concentration of durvalumab at steady state is reported.
Trough Concentration at Steady State (Ctrough) of Durvalumab | Cohorts A and B: Pre-dose on Day 141; Cohort C: Pre-dose on Day 169
  Trough concentration of durvalumab pre-dose at steady state is reported.
Number of Participants With Postive Anti-Drug Antibodies (ADA) Titer to Durvalumab | Cohorts A and B: Days 1 and 29; Cohort C: Days 29 and 57
  The number of participants with positive serum antibodies to durvalumab post dosing are reported.

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — MedImmune LLC
Locations (11):
- United States (7):
  - Research Site, Scottsdale, Arizona
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Miami Beach, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Villejuif, France
- Research Site, Napoli, Italy

REFERENCES:
- [Background] Gordon MS, Lutzky J, Lawrence D, Butler M, Ascierto PA, Hug B, et al. Phase 1 study evaluating safety and tolerability of MEDI4736, an anti-programmed cell death ligand-1 (PD-L1) antibody, in combination with dabrafenib and trametinib or trametinib alone in patients with unresectable or metastatic melanoma. Ann Oncol 2014; 25(suppl_4): iv374-iv393 (abstract 8004).
- [Result] Ribas A, Butler M, Lutzky J, Lawrence DP, Robert C, Miller W, et al. Phase 1 study combining anti-PD-L1 (MEDI4736) and BRAF (dabrafenib) and/or MEK (trametinib) inhibitors in advanced melanoma. J Clin Oncol 2015; 33 (15_suppl): (abstract 3003).
- [Derived] Ribas A, Algazi A, Ascierto PA, Butler MO, Chandra S, Gordon M, Hernandez-Aya L, Lawrence D, Lutzky J, Miller WH Jr, Campbell KM, Delafont B, Marshall S, Mueller N, Robert C. PD-L1 blockade in combination with inhibition of MAPK oncogenic signaling in patients with advanced melanoma. Nat Commun. 2020 Dec 7;11(1):6262. doi: 10.1038/s41467-020-19810-w. PMID 33288749